CLINICAL TRIAL: NCT04265417
Title: Clinical Outcomes and Prognostic Factors of Robotic Assisted Rectal Cancer Resection Alone vs. Robotic Rectal Cancer Resection With Natural Orifice Specimen Extraction
Status: Completed | Type: Observational
Sponsor: Taiyuan Li (Other)
Responsible Party: Sponsor-Investigator, Taiyuan Li, Prof., Chief physician, Head of The Fifth Department of General Surgery, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Other Study IDs: RARN
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Rectal Neoplasms; Robotic Surgery; Natural Orifice Specimen Extraction Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The resected specimens were kept and sent to the laboratory for pathological examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RARC group: Participants in this group underwent robotic assisted rectal cancer resection
  Interventions: Procedure: Robotic Assisted Rectal Cancer Resection Alone
- NOSE group: Participants in this group underwent robotic rectal cancer resection assisted rectal with natural orifice extraction
  Interventions: Procedure: Robotic Assisted Rectal Cancer Resection With Natural Orifice Specimen Extraction

INTERVENTIONS:
Procedure: Robotic Assisted Rectal Cancer Resection Alone — participants in this group underwent robotic assisted rectal cancer resection alone, the specimens were extracted through the incision on the abdominal wall.
  Groups: RARC group
Procedure: Robotic Assisted Rectal Cancer Resection With Natural Orifice Specimen Extraction — participants in this group underwent robotic rectal cancer resection，the specimens were extractd through anus and vagina.
  Groups: NOSE group

SUMMARY:
Robotic rectal cancer resection with natural orifice extraction is a recently developed minimally invasive surgery for patients with rectal cancer. However, it's safety and feasibility remain undiscussed and controversial. This study reported the clinical outcomes and prognostic factors of robotic assisted rectal cancer resection alone vs. robotic rectal cancer resection with natural orifice extraction to discuss aforementioned question.

DETAILED DESCRIPTION:
Robotic rectal cancer resection with natural orifice extraction is a recently developed minimally invasive surgery for patients with rectal cancer. However, it's safety and feasibility remain undiscussed and controversial. This study reported the clinical outcomes and prognostic factors of robotic assisted rectal cancer resection alone vs. robotic rectal cancer resection with natural orifice extraction to discuss aforementioned question. From January 2015 to November 2016, a consecutive wave of 49 patients underwent robotic rectal cancer resection with natural orifice extraction and 49 matched patients underwent conventional robotic assisted rectal cancer resection were systematically analyzed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. T stage 1-3;
2. aged between 18 to 75;
3. the tumor margin is at least 4 cm from the anus;
4. body mass index ≤30kg/m2;
5. no distant metastases； (6）tumor size≤5cm.

Exclusion Criteria:

1. emergency surgery for intestinal obstruction or massive bleeding;
2. history of abdominal or pelvic surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2015 to November 2016, a consecutive wave of patients with rectal cancer underwent conventional robotic assisted rectal cancer resection and robotic rectal cancer resection with natural orifice extraction were invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 36 months
  To determine the survival differences between NOSE group and RARC group. Overall survival is defined as the time from surgery to death from any causes
Disease-free survival | Up to 36 months
  To determine the survival differences between NOSE group and RARC group. Disease-free survival is defined as the time from surgery to local or distant recurrence

SECONDARY OUTCOMES:
Operation time | 1 day
  To determine the differences between NOSE group and RARC group
Estimated intraoperative blood loss | 1 day
  To determine the differences between NOSE group and RARC group
Postoperative hospital stay | 30 days
  To determine the surgical and patients burdern differences between NOSE group and RARC group
Postoperative visual analogue scale scale on day 1 | 1 day
  To determine the surgical differences between NOSE group and RARC group. Maxium sacle is 10, miniun scale is 0. 0 represents no pain. 10 represents maximun pain.
Time to pass flatus | 30 days
  To determine the surgical differences between NOSE group and RARC group
Hospitalization costs | 30 day
  to determine the patients burden differences between NOSE group and RARC group
Specimen length | 30 day
  To determine the surgical differences between NOSE group and RARC group
Proximal margin | 30 day
  To determine the pathological differences between NOSE group and RARC group
Distal margin | 30 days
  To determine the pathological differences between NOSE group and RARC group
Histological differentiation | 30 days
  To determine the pathological differences between NOSE group and RARC group
Number of lymph nodes harvested | 30 days
  To determine the pathological differences between NOSE group and RARC group
Postoperative white blood cell count | 30 days
  To determine the surgical stress response differences NOSE group and RARC group
Postoperative procalcitonin | 30 days
  To determine the surgical stress response differences NOSE group and RARC group
Postoperative C-reactive protein | 30 days
  To determine the surgical stress response differences NOSE group and RARC group

IPD SHARING:
Plan to Share IPD: No